CLINICAL TRIAL: NCT04713787
Title: A Phase 2, Partially-Blinded, Randomized, Comparative Study of the Efficacy of Different Doses of Oxfendazole Compared to a Single Dose of Albendazole for the Treatment of Trichuris Trichiura Infection in Adults
Brief Title: A Safety and Efficacy Study of Different Doses of Oxfendazole Compared to a Single Dose of Albendazole to Treat Trichuris Trichiura Infection in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asociacion Benefica Prisma (Other)
Collaborators: Policlinico Asociacion Benefica PRISMA-Laboratorio Satelite IQTLAB (Unknown); National Institutes of Health (NIH) (NIH); University of Iowa (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0004; HHSN272201300020I; IND158335 (Other: FDA)
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Trichuriasis
Keywords: Adults; Albendazole; Comparative Study; Efficacy; Oxfendazole; Phase 2; Trichuris trichiura
MeSH Terms: conditions — Trichuriasis | interventions — Albendazole; oxfendazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is masked only to the laboratory personnel. All stool samples, labelled only with a barcode and the date of sample collection by the study team will be evaluated by blinded laboratory staff and will remain blinded until locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): 400 mg (4 capsules of 100 mg) of Oxfendazole administered orally as a single dose on Day 1. N=83.
  Interventions: Drug: Oxfendazole
- Group B (Experimental): 800 mg (8 capsules of 100 mg) of Oxfendazole administered orally as a single dose on Day 1. N=83.
  Interventions: Drug: Oxfendazole
- Group C (Active Comparator): 400 mg (1 tablet of 400 mg) of Albendazole administered orally as a single dose on Day 1. N=83.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — Albendazole, 5-(prophylthio)-2-benzimidazole carbamate, is a broad-spectrum benzimidazole antihelminthic drug. It is provided as a white to off-white, circular, film-coated tablet with a slightly raised pentagonal projection on either side. This trial will use the 400 mg tablet formulation.
  Arms: Group C
Drug: Oxfendazole — The active pharmaceutical ingredient is methyl-5 (6)-phenylsulfiyl-2-benzimidazole carbamate, which is a broad-spectrum benzimidazole antihelminthic. Oxfendazole is the sulphoxide metabolite of fenbendazole.
  Arms: Group A; Group B

SUMMARY:
This is a Phase 2 trial to evaluate the efficacy of different doses of oxfendazole versus a single dose of albendazole in curing or reducing the egg burden in subjects with T. trichiura infections. 249 subjects will be randomized in a 1:1:1 ratio to one of three dose-groups to receive a single dose of oxfendazole 400 mg or 800 mg, or a single dose of albendazole 400 mg. The study team members and study subjects will not be blinded to the dose group. However, the laboratory assessors evaluating the stool samples will be blinded. Subjects will be recruited in Iquitos, Peru, and surrounding villages where there is a high prevalence of T. trichiura infection. Subjects will be solicited through town hall meetings and local clinics and through recommendations from local care providers. A two-stage screening process will be utilized. If subjects are found on the screening stool exam to have only a stool parasite other than T. trichuria or if the subject chooses not to participate in the study, the subject will be referred to a local health provider. If stool analysis performed at the end of the study period demonstrates stool parasites, the subjects will be contacted and referred to their local health provider where they will receive standard of care treatment. The primary objective is to assess the cure rate of different dose regimens of oxfendazole vs. albendazole in the treatment of T. trichiura infections using the Kato-Katz stool examination method.

DETAILED DESCRIPTION:
This is a Phase 2 trial to evaluate the efficacy of different doses of oxfendazole versus a single dose of albendazole in curing or reducing the egg burden in subjects with T. trichiura infections. 249 subjects will be randomized in a 1:1:1 ratio to one of three dose-groups to receive a single dose of oxfendazole 400 mg or 800 mg, or a single dose of albendazole 400 mg. Water and a snack will be provided to aid in ingestion of the study product and a study team member will observe the ingestion of study product. The study team members and study subjects will not be blinded to the dose group. However, the laboratory assessors evaluating the stool samples will be blinded. Subjects will be recruited in Iquitos, Peru, and surrounding villages where there is a high prevalence of T. trichiura infection. Subjects will be solicited through town hall meetings and local clinics and through recommendations from local care providers. A two-stage screening process will be utilized. If subjects are found on the screening stool exam to have only a stool parasite other than T. trichuria or if the subject chooses not to participate in the study, the subject will be referred to a local health provider. If stool analysis performed at the end of the study period demonstrates stool parasites, the subjects will be contacted and referred to their local health provider where they will receive standard of care treatment. The primary objective is to assess the cure rate of different dose regimens of oxfendazole vs. albendazole in the treatment of T. trichiura infections using the Kato-Katz stool examination method. The secondary objectives are to: 1) assess the cure rate of different dose regimens of oxfendazole vs albendazole in the treatment of T. trichiura infections using the stool concentration examination method, 2) assess the clinical response compared to baseline, as shown by reduction in T. trichiura egg counts using the Kato-Katz stool examination method, 3) assess the clinical response compared to baseline, as shown by reduction in T. trichiura egg counts using the stool concentration method, 4) assess the proportion of subjects with moderate or heavy infection before treatment who had no infection or only light infection after treatment using the Kato-Katz stool examination method, 5) assess the proportion of subjects with moderate or heavy infection before treatment who had no infection or only light infection after treatment using the stool concentration examination method, 6) establish the spectrum of activity of oxfendazole against other intestinal helminths using the Kato-Katz stool examination method, 7) establish the spectrum of activity of oxfendazole against other intestinal helminths using the stool concentration examination method, 8) assess the tolerability of each oxfendazole dose group compared to the albendazole dose group, and 9) assess the safety in subjects treated with oxfendazole.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-65 years, inclusive and weigh ≥45 kg.
2. Are willing to participate in this trial, as evidenced by written or witnessed oral informed consent.
3. T. trichiura* is demonstrated in a stool sample obtained within 14 days before randomization and enrollment.

   *The presence of A. lumbricoides, N. americanus, A. duodenalis, or other helminths will not be a cause for exclusion.
4. Are willing to comply with the requirements of this protocol, particularly to provide four stool samples and two blood samples* over approximately 4- 6 weeks.

   *An extra stool or blood sample might be required if the samples are not collected within the appropriate time frame or to follow up on abnormal laboratory tests.
5. Females must have a negative serum pregnancy test within 10 days or a negative urine pregnancy test 72 hours prior to the first study drug administration.*ª

   *If a woman of child bearing potential is on an injectable form of contraception, a single serum pregnancy test at screening (Days -10 to -1) is acceptable. If the woman is not using an injectable form of contraception, a pregnancy test must be negative 72 hours prior to the first study drug administration.

   ª Pregnancy testing is not required for women of non-childbearing potential
6. Female subjects of childbearing potential must be using effective contraception.* *Effective methods of contraception include: abstinence from sexual intercourse, monogamous relationship with a vasectomized partner, male condoms with spermicide, surgical sterility, intrauterine contraceptive device, oral or injectable contraceptives, diaphragm in combination with contraceptive cream or foam. Females aged >/=50 years who have had no menstrual periods for 1 year may be enrolled. Females must agree to continue effective contraception for approximately 28 days following the last study drug administration.

Exclusion Criteria:

1. Has demonstrated a previous hypersensitivity reaction to oxfendazole or a related compound (e.g. albendazole, mebendazole).
2. Has a diarrheal disease that would interfere with the evaluation of stool samples*.

   * More than 6 stools per day or stools that are completely liquid.
3. Has received an antihelminthic within 14 days before enrolment.
4. Has received an investigational drug within 30 days before the screening visit or is scheduled to receive such a drug during this trial.
5. Has a concomitant infection or another underlying disease that would compromise the safety, diagnosis, and evaluation of responses to the study drug.
6. Has a known history of renal dysfunction or plasma creatinine >/=1.5 times the upper limit of normal (ULN) for age.
7. Has a known history of hepatic dysfunction or AST, ALT, total bilirubin >/=1.5 times the ULN.
8. Has a hemoglobin that is less than 8 g/dL.
9. Is a female who is pregnant, lactating, or planning a pregnancy during this trial (up to days 28 after the last scheduled dose).
10. Has previously been enrolled in this trial.
11. Has any condition that would, in the investigator's opinion, interfere with this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of infection cures (Clinical Cure) as shown by absence of Trichuris trichiura eggs using the Kato-Katz stool examination method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from two stools samples (each evaluated in duplicate).

SECONDARY OUTCOMES:
Change from baseline in eggs per gram of stool for helminths other than Trichuris trichiura using the Kato Katz examination method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from two stools samples (each evaluated in duplicate).
Change from baseline in eggs per gram of stool for helminths other than Trichuris trichiura using the stool concentration examination method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from two stools samples (each evaluated in duplicate).
Change from baseline in eggs per gram of stool using the Kato-Katz stool examination method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from two stools samples (each evaluated in duplicate).
Change from baseline in eggs per gram of stool using the stool concentration method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from two stools samples (each evaluated in duplicate).
Egg reduction rate, relative to egg counts at baseline, measured using the Kato-Katz stool examination method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from egg counts (eggs per gram) from two stool samples (each evaluated in duplicate).
Egg reduction rate, relative to egg counts at baseline, using the stool concentration method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from egg counts (eggs per gram) from two stool samples (each evaluated in duplicate).
Number of infection cures (Clinical Cure) as shown by absence of Trichuris trichiura eggs using the stool concentration method | Day 18 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Calculated from two stools samples (each evaluated in duplicate).
Proportion of abnormal laboratory tests | Day 1 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Abnormal laboratory tests include hemoglobin (Hgb), white blood cells (WBC), neutrophil and eosinophil counts, platelet counts, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, alkaline phosphatase, and creatinine.
Proportion of solicited clinical reactogenicity events | Day 1 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group. Solicited clinical reactogenicity events including nausea, vomiting, abdominal pain, diarrhea, and anorexia.
Proportion of subjects in each dose group with moderate or heavy infection who had no infection or only light infection after treatment based on WHO classes of intensity, measured using the Kato-Katz tool examination method | Day 18 through Day 23
  According to WHO thresholds, infections of 1-999 eggs per gram (epg) are classified as light intensity infections, 1,000-9,999 epg are classified as moderate, and >/= 10,000 epg are classified as heavy.
  Classification at baseline will be based on the screening stool sample, and classification post-treatment will be based on two stool samples each oxfendazole dose group compared to the albendazole dose group.
Proportion of unsolicited adverse events (AEs) | Day 1 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group.
Serious adverse events (SAEs) related to the study product | Day 1 through Day 23
  As measured in each oxfendazole dose group compared to the albendazole dose group.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Asociacion Benefica Prisma, Santa Clara de Nanay, Maynas, Peru

IPD SHARING:
Plan to Share IPD: Undecided